CLINICAL TRIAL: NCT01903941
Title: Anti-inflammatory Effect of Aerobic Exercise in Individual With Increased Cardiovascular Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Escola Bahiana de Medicina e Saude Publica (Other)
Responsible Party: Principal Investigator, Luis CL Correia, Associate Professor of Medicine, Escola Bahiana de Medicina e Saude Publica
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRPExercise
Record Dates: First submitted 2013-06-28; First posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Inflammation
Keywords: exercise
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training (Experimental): Aerobic
  Interventions: Behavioral: Aerobic Exercise
- Control (Placebo Comparator): Not exercise
  Interventions: Behavioral: Only Counseling

INTERVENTIONS:
Behavioral: Aerobic Exercise
  Arms: Training
Behavioral: Only Counseling
  Arms: Control

SUMMARY:
Aerobic physical activity attenuates systemic inflammatory activity in individuals with cardiovascular risk.

DETAILED DESCRIPTION:
Background: Observational studies suggest that exercise has anti-inflammatory effect, however this idea has not been definitively confirmed by randomized clinical trials.

Objective: To test the hypothesis that aerobic exercise attenuates systemic inflammatory activity in individuals with cardiovascular risk.

Methods: Randomized controlled trial, which included 68 sedentary individuals, with at least two risk factors for coronary heart disease or established cardiovascular disease. The volunteers were randomized to 3 months of supervised aerobic training or just advice when healthy lifestyles. C-reactive protein (CRP) was measured by the method of high sensitivity before and after 3 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

- Individuals with are between 40 to 70 years, no regular exercise, and at least two risk factor for cardiovascular disease (diabetes, hypertension, dyslipidemia, smoking) or documented cardiovascular disease.

Exclusion Criteria:

- Incapacity to exercise.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2006-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | 3 months